CLINICAL TRIAL: NCT00819156
Title: An Open-label, Randomised, Multi-centre, Parallel Group Comparison of the Efficacy and Safety of Degarelix at Six Different Dosing Regimens in Patients With Prostate Cancer Treated for 12 Months
Brief Title: Dose Finding Trial With a New Treatment (Degarelix) for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS12
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2011-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Degarelix 200/80 (Experimental): Cycle 1 was an initial 200 milligram dose of Degarelix. Cycles 2-13 were maintenance doses of 80 milligrams each of Degarelix. Each cycle was 28 days.
  Interventions: Drug: degarelix
- Degarelix 200/120 (Experimental): Cycle 1 was an initial 200 milligram dose of Degarelix. Cycles 2-13 were maintenance doses of 120 milligrams each of Degarelix. Each cycle was 28 days.
  Interventions: Drug: degarelix
- Degarelix 200/160 (Experimental): Cycle 1 was an initial 200 milligram dose of Degarelix. Cycles 2-13 were maintenance doses of 160 milligrams each of Degarelix. Each cycle was 28 days.
  Interventions: Drug: degarelix
- Degarelix 240/80 (Experimental): Cycle 1 was an initial 240 milligram dose of Degarelix. Cycles 2-13 were maintenance doses of 80 milligrams each of Degarelix. Each cycle was 28 days.
  Interventions: Drug: degarelix
- Degarelix 240/120 (Experimental): Cycle 1 was an initial 240 milligram dose of Degarelix. Cycles 2-13 were maintenance doses of 120 milligrams each of Degarelix. Each cycle was 28 days.
  Interventions: Drug: degarelix
- Degarelix 240/160 (Experimental): Cycle 1 was an initial 240 milligram dose of Degarelix. Cycles 2-13 were maintenance doses of 160 milligrams each of Degarelix. Each cycle was 28 days.
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix — Degarelix was given as subcutaneous injections.
  Other Names: FE200486

SUMMARY:
The purpose of the trial was to evaluate the safety and efficacy of degarelix when comparing six different doses. The patients participating in the trial were treated with degarelix every month for a year. During the treatment the patients had to visit the clinic for investigations. Blood samples for testosterone, dihydrotestosterone, luteinizing hormone, follicle stimulating hormone, and Prostate Specific Antigen were taken and analysed throughout the trial.

DETAILED DESCRIPTION:
Degarelix was not FDA regulated at the time of the trial. After completion of the trial degarelix has been approved by the FDA and is thus an FDA regulated intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study related procedures
* Proven prostate cancer in need for endocrine treatment, except for neoadjuvant hormonal therapy, but including patients with a rising PSA further to prostatectomy or radiotherapy
* ECOG score to be equal to or above 2
* Testosterone level within age-specific normal range
* PSA value equal to or above 2 ng/ml
* Life expectancy of at least 6 months

Exclusion Criteria:

* Previous or current hormonal treatment of prostate cancer
* Recent or current treatment with any drugs modifying the testosterone level
* Candidate for curative treatment such as prostatectomy or radiotherapy
* History of severe asthma, anaphylactic reactions, angioedema, angioneurotic oedema or Quincke's Oedema
* Hypersensitivity towards any component of degarelix or mannitol
* Cancer disease within the last 5 years except for prostate cancer and some skin cancers
* Signs of liver impairment shown as elevated serum ALT or serum bilirubin
* Known hepatic disease
* Other laboratory abnormalities that judged by the investigator would interfere with the patients participation in the trial or the evaluation of the trial results
* Clinically significant disorder including excessive alcohol or drug abuse that may interfere with trial participation or influence the conclusion of the trial as judged by the investigator
* Mental incapacity or language barrier precluding adequate understanding or cooperation
* Having received an investigational product within the last 12 weeks preceding the trial
* Previous participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2004-02; Primary Completion 2005-06 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (39):
- Belgium (3):
  - UCL Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Germany (4):
  - Vivantes Klinikum am Urban, Berlin
  - Loretto Krankenhaus, Freiburg im Breisgau
  - Euromed AG Klinik, Fürth
  - Urologische Universitätsklinikum, Mannheim
- Hungary (6):
  - Bajcsy-Zsilinszky Hospital, Urology, Budapest
  - Jahn Ferenc Dél Pesti Hospital, Urology, Budapest
  - Pez Aladar County Hospital, Győr
  - BAZ County Hospital, Miskolc
  - Hospital of Local Gov. Szeged, Urology, Szeged
  - MÁV Hospital, Urology, Szolnok
- Netherlands (2):
  - AMC, Amsterdam
  - Atrium MC, Heerlen
- Poland (2):
  - Wojewódzki Szpital Specjalisttyczny, Siedlce
  - Wojewódzki Szpital Specjalisttyczny, Słupsk
- Romania (4):
  - CF2 Hospital, Bucharest
  - Dr. Th Burghele Hospital, Bucharest
  - Fundeni Hospital, Bucharest
  - Sf. Ioan Hospital, Bucharest
- Russia (13):
  - Botkin Clinical Hospital, Moscow
  - City Hospital #1, Moscow
  - City Hospital #29, Moscow
  - City Hospital #50, Moscow
  - City Hospital #60, Moscow
  - Institute of Urology of MoH, Moscow
  - "Andros" Urology Clinic, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - Military Medical Academy, Urology, Saint Petersburg
  - Pavlov Medical School Outpatient, Saint Petersburg
  - Pavlov medical School, Urology, Saint Petersburg
  - Sct Petersburg State Medical Academy, Saint Petersburg
- South Africa (5):
  - 370 Clarke Road, Glenwood, Durban
  - Pretoria Urology Hospital, Hatfield, Pretoria
  - WITS Medical School, Parktown
  - 401B Medical Centre, Pietermaritzburg
  - Sunninghill Clinic, Sunninghill

REFERENCES:
- [Result] Van Poppel H, Tombal B, de la Rosette JJ, Persson BE, Jensen JK, Kold Olesen T. Degarelix: a novel gonadotropin-releasing hormone (GnRH) receptor blocker--results from a 1-yr, multicentre, randomised, phase 2 dosage-finding study in the treatment of prostate cancer. Eur Urol. 2008 Oct;54(4):805-13. doi: 10.1016/j.eururo.2008.04.065. Epub 2008 May 8. PMID 18538469

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred and sixteen patients were screened. Twenty-seven were screening failures. Two randomized patients were not treated: one withdrew consent and the other had an elevated alanine aminotransferase value (an exclusion criteria found after randomization).
Groups:
- Degarelix 200/80: Cycle 1 was an initial 200 milligram dose of Degarelix. Cycles 2-13 were maintainance doses of 80 milligrams each of Degarelix. Each cycle was 28 days.
- Degarelix 200/120: Cycle 1 was an initial 200 milligram dose of Degarelix. Cycles 2-13 were maintainance doses of 120 milligrams each of Degarelix. Each cycle was 28 days.
- Degarelix 200/160: Cycle 1 was an initial 200 milligram dose of Degarelix. Cycles 2-13 were maintainance doses of 160 milligrams each of Degarelix. Each cycle was 28 days.
- Degarelix 240/80: Cycle 1 was an initial 240 milligram dose of Degarelix. Cycles 2-13 were maintainance doses of 80 milligrams each of Degarelix. Each cycle was 28 days.
- Degarelix 240/120: Cycle 1 was an initial 240 milligram dose of Degarelix. Cycles 2-13 were maintainance doses of 120 milligrams each of Degarelix. Each cycle was 28 days.
- Degarelix 240/160: Cycle 1 was an initial 240 milligram dose of Degarelix. Cycles 2-13 were maintainance doses of 160 milligrams each of Degarelix. Each cycle was 28 days.
Period: Overall Study
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Started | 30 | 33 | 32 | 30 | 33 | 31
Randomised and Treated (ITT Population) | 30 | 32 | 32 | 30 | 33 | 30
Completed | 20 | 23 | 26 | 28 | 27 | 23
Not Completed | 10 | 10 | 6 | 2 | 6 | 8
Not completed — Adverse Event | 1 | 4 | 2 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Testosterone >1ng/ml from Day 28+ | 5 | 2 | 1 | 1 | 1 | 2
Not completed — Testosterone >=.5ng/ml 2 visits | 3 | 0 | 0 | 0 | 1 | 0
Not completed — Prostate-specific antigen progression | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160 | Total
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 5 | 6 | 7 | 7 | 37
  >=65 years | 23 | 27 | 27 | 24 | 26 | 23 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.27) | 70.6 (7.72) | 73.3 (7.39) | 70.4 (7.07) | 70.7 (7.56) | 70.7 (8.59) | 70.9 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 30 | 32 | 32 | 30 | 33 | 30 | 187
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 2 | 0 | 6
  White | 29 | 30 | 31 | 30 | 30 | 30 | 180
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Number of Patients at Each Stage of Prostate Cancer [Number; unit: patients] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tummors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  patients
    Localized | 8 | 6 | 6 | 5 | 11 | 5 | 41
    Locally advanced | 8 | 11 | 11 | 12 | 8 | 10 | 60
    Metastatic | 4 | 8 | 5 | 5 | 7 | 7 | 36
    Not classifiable | 10 | 7 | 10 | 8 | 7 | 8 | 50
Patient Counts by Gleason Score [Number; unit: participants] — The Gleason Score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10 with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    unknown | 0 | 0 | 2 | 0 | 0 | 0 | 2
    2-4 | 4 | 10 | 6 | 9 | 4 | 3 | 36
    5-6 | 13 | 10 | 14 | 10 | 17 | 12 | 76
    7-10 | 13 | 12 | 10 | 11 | 12 | 15 | 73
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] — Body mass index is a measure of body fat based on height and weight.
  kilograms per square meter | 26.4 (3.5) [18.1 to 36] | 26.4 (3.74) [20.3 to 36.8] | 25.9 (4.46) [17.9 to 36.3] | 27.7 (5.3) [18.5 to 41.1] | 26 (3.28) [18.2 to 32.7] | 25.3 (2.73) [20.3 to 29.8] | 26.3 (3.94) [17.9 to 41.1]
Days Since Diagnosis of Prostate Cancer [Mean (Standard Deviation); unit: days] — The mean number of days that have passed since a diagnosis of prostate cancer was made for each patient.
  days | 493 (849) | 122 (230) | 375 (1098) | 383 (817) | 229 (508) | 352 (743) | 323 (756)
Median Serum Testosterone Level [Median (Full Range); unit: nanogram / milliliter] — Testosterone is a steroid hormone from the androgen group, and the principal male sex hormone. This test measures the amount of testosterone in the blood. Androgen deprivation is used to manage prostate cancer.
  nanogram / milliliter | 4.47 [0.816 to 7.1] | 3.93 [1.53 to 9.29] | 4.79 [2.8 to 9.47] | 4.28 [1.4 to 10.2] | 4.07 [2.02 to 7.7] | 3.88 [1.69 to 8.63] | 4.13 [0.816 to 10.2]
Serum Prostate-specific Antigen [Median (Full Range); unit: nanogram / milliliter] — Prostate-specific antigen (PSA) is a protein produced by the cells of the prostate gland. The PSA test measures the level of PSA in the blood. High PSA levels have a positive correlation to prostate cancer.
  nanogram / milliliter | 15.2 [2.6 to 332] | 31.5 [3.3 to 1730] | 31.5 [2.6 to 901] | 23.1 [3.6 to 586] | 35.3 [2.4 to 1110] | 32 [2 to 1297] | 27.6 [2 to 1730]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Testosterone <=0.5 Nanograms/Milliliter From Day 28 to Day 364
Description: Number of patients who achieved a testosterone level considered a castration level.
Time Frame: 12 months
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 28 | 25 | 27 | 30 | 30 | 25
participants | 17 [41 to 78] | 21 [64 to 95] | 26 [81 to 100] | 27 [73 to 98] | 27 [73 to 98] | 23 [74 to 99]
Statistical Analysis 1: Comparison: Degarelix 200/80; Test type: Superiority or Other; Percentage = 61, 95% CI [41 to 78] — The estimated value is the percentage of patients with Testosterone <=0.5 nanograms/milliliter from Day 28 to Day 364. The 95% Confidence Interval was calculated by the Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 200/120; Test type: Superiority or Other; Percentage = 84, 95% CI [64 to 95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Degarelix 200/160; Test type: Superiority or Other; Percentage = 96, 95% CI [81 to 100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Degarelix 240/80; Test type: Superiority or Other; Percentage = 90, 95% CI [73 to 98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Degarelix 240/120; Test type: Superiority or Other; Percentage = 90, 95% CI [73 to 98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Degarelix 240/160; Test type: Superiority or Other; Percentage = 92, 95% CI [74 to 99] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Patients With Testosterone Level <=0.5 Nanogram/Milliliter From Day 28 to Day 364 for Patients With Testosterone <=0.5 Nanogram/Milliliter at Day 28
Description: Number of patients who maintained a castration level of testosterone (<=0.5 Nanogram/Milliliter) while on a maintenance dose of Degarelix from Day 28 - 364.
Time Frame: Day 28 - 364
Population: ITT population of patients with testoterone measurements <=0.5 nanogram/milliliter at Day 28.
Measure: Number; unit: participants
Groups:
- Maintenance Dose of 80 Milligram Per Cycle: The two treatment groups that have a maintenance dose of 80 milligram per cycle in cycles 2-13 have been combined.
- Maintenance Dose of 120 Milligram Per Cycle: The two treatment groups that have a maintenance dose of 120 milligram per cycle in cycles 2-13 have been combined.
- Maintenance Dose of 160 Milligram Per Cycle: The two treatment groups that have a maintenance dose of 160 milligram per cycle in cycles 2-13 have been combined.
Arm/Group | Maintenance Dose of 80 Milligram Per Cycle | Maintenance Dose of 120 Milligram Per Cycle | Maintenance Dose of 160 Milligram Per Cycle
Number analyzed (Participants) | 48 | 50 | 49
participants | 44 [80 to 98] | 48 [86 to 100] | 49 [93 to 100]
Statistical Analysis 1: Comparison: Maintenance Dose of 80 Milligram Per Cycle; Test type: Superiority or Other; Percentage = 92, 95% CI [80 to 98] — The estimated value is the percentage of patients with Testosterone (T) <=0.5 nanograms (ng)/milliliter (mL) from Day 28 to Day 364 for Patients With T <=0.5 ng/mL at Day 28. The 95% Confidence Interval was calculated by the Clopper-Pearson method
Statistical Analysis 2: Comparison: Maintenance Dose of 120 Milligram Per Cycle; Test type: Superiority or Other; Percentage = 96, 95% CI [86 to 100] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Maintenance Dose of 160 Milligram Per Cycle; Test type: Superiority or Other; Percentage = 100, 95% CI [93 to 100] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Patients With Testosterone <=0.5 Nanogram/Milliliter at Day 28.
Description: The number of patients who achieved the <=0.5 nanogram/milliliter level for serum testosterone after the initial dose cycle.
Time Frame: Day 28
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
participants | 21 [51 to 85] | 29 [75 to 98] | 31 [84 to 100] | 29 [83 to 100] | 31 [80 to 99] | 27 [77 to 99]
Statistical Analysis 1: Comparison: Degarelix 200/80; Test type: Superiority or Other; Percentage = 70, 95% CI [51 to 85] — The estimated value is the percentage of patients with Testosterone <=0.5 nanograms/milliliter at Day 28. The 95% Confidence Interval was calculated with the Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 200/120; Test type: Superiority or Other; Percentage = 91, 95% CI [75 to 98] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Degarelix 200/160; Test type: Superiority or Other; Percentage = 97, 95% CI [84 to 100] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Degarelix 240/80; Test type: Superiority or Other; Percentage = 97, 95% CI [83 to 100] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Degarelix 240/120; Test type: Superiority or Other; Percentage = 94, 95% CI [80 to 99] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Degarelix 240/160; Test type: Superiority or Other; Percentage = 93, 95% CI [77 to 99] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Number of Patients With Testoterone <=0.5 Nanogram/Milliliter at Day 3.
Description: The number of patients who achieved the <=0.5 nanogram/milliliter level for serum testosterone after 3 days.
Time Frame: Day 3
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
participants | 25 [65 to 94] | 30 [79 to 99] | 27 [70 to 96] | 28 [78 to 99] | 30 [76 to 98] | 28 [78 to 99]
Statistical Analysis 1: Comparison: Degarelix 200/80; Test type: Superiority or Other; Percentage = 83, 95% CI [65 to 94] — The estimated value is the percentage of patients with Testosterone <=0.5 nanograms/milliliter at Day 3. The 95% Confidence Interval was calculated with the Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 200/120; Test type: Superiority or Other; Percentage = 94, 95% CI [79 to 99] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Degarelix 200/160; Test type: Superiority or Other; Percentage = 87, 95% CI [70 to 96] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Degarelix 240/80; Test type: Superiority or Other; Percentage = 93, 95% CI [78 to 99] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Degarelix 240/120; Test type: Superiority or Other; Percentage = 91, 95% CI [76 to 98] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Degarelix 240/160; Test type: Superiority or Other; Percentage = 93, 95% CI [78 to 99] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Days to 50 Percent Reduction in Prostate-Specific Antigen
Description: Median number of days after the first dose of Degarelix when the prostate-specific antigen levels fell to 50 percent of the baseline value.
Time Frame: Day 0 (post dose) to Day 364
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
days | 14 [7 to 224] | 14 [3 to 84] | 14 [3 to 42] | 14 [3 to 56] | 14 [3 to 84] | 14 [3 to 56]
Statistical Analysis 1: Comparison: Degarelix 200/80 vs Degarelix 200/120 vs Degarelix 200/160 vs Degarelix 240/80 vs Degarelix 240/120 vs Degarelix 240/160; Test type: Superiority or Other; p = 0.0933, Log Rank

6. Secondary Outcome: Days to 90 Percent Reduction in Prostate-Specific Antigen
Description: Median number of days after the first dose of Degarelix when the prostate-specific antigen levels fell to 90 percent of the baseline value.
Time Frame: Day 0 (post dose) to Day 364
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
days | 56 [28 to 168] | 56 [14 to 336] | 56 [14 to 336] | 56 [14 to 196] | 56 [28 to 364] | 56 [14 to 196]
Statistical Analysis 1: Comparison: Degarelix 200/80 vs Degarelix 200/120 vs Degarelix 200/160 vs Degarelix 240/80 vs Degarelix 240/120 vs Degarelix 240/160; Test type: Superiority or Other; p = 0.165, Log Rank

7. Secondary Outcome: Days to Prostate-Specific Antigen Progression
Description: Median days to prostate-specific antigen increase of >= 50 percent and >=5 nanograms/milliliter compared to nadir on two consecutive visits at least two weeks apart.
Time Frame: Day 0 (post dose) to Day 364
Population: Number of patients with PSA progression in the six groups n=0,3,1,4,4,2. Since no patients in the 200/80 group experience PSA progression the Days to progression could not be calculated.
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 32 | 32 | 30 | 33 | 30
days | 224 [140 to 308] | 308 [308 to 308] | 280 [252 to 336] | 224 [126 to 364] | 140 [140 to 140]
Statistical Analysis 1: Comparison: Degarelix 200/120 vs Degarelix 200/160 vs Degarelix 240/80 vs Degarelix 240/120 vs Degarelix 240/160; Test type: Superiority or Other; p = 0.429, Log Rank

8. Secondary Outcome: Median Serum Testosterone Levels
Time Frame: Day 0 (Baseline), Days 1,3,7,14, and 364
Population: ITT population
Measure: Median (Full Range); unit: nanogram/milliliter
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
nanogram/milliliter
  Day 0 (Baseline) | 4.47 [0.816 to 7.1] | 3.93 [1.53 to 9.29] | 4.79 [2.8 to 9.47] | 4.28 [1.4 to 10.2] | 4.07 [2.02 to 7.7] | 3.88 [1.69 to 8.63]
  Day 1 (n=30,32,32,30,33,30) | 0.654 [0.167 to 1.81] | 0.436 [0.207 to 1.21] | 0.465 [0.287 to 2.44] | 0.563 [0.2 to 3] | 0.453 [0.21 to 3.32] | 0.576 [0.261 to 1.36]
  Day 3 (n=30,32,31,30,33,30) | 0.308 [0.121 to 2.81] | 0.26 [0.139 to 0.657] | 0.281 [0.125 to 0.64] | 0.265 [0.119 to 0.586] | 0.268 [0.133 to 0.912] | 0.261 [0.144 to 1.3]
  Day 7 (n=30,32,32,30,33,28) | 0.283 [0.098 to 4] | 0.237 [0.066 to 1.43] | 0.198 [0.087 to 0.808] | 0.193 [0.104 to 0.549] | 0.216 [0.116 to 1.55] | 0.207 [0.074 to 4.66]
  Day 14 (n=30,32,32,30,33,29) | 0.173 [0.025 to 4.77] | 0.144 [0.054 to 1.62] | 0.122 [0.025 to 0.617] | 0.152 [0.025 to 0.641] | 0.134 [0.05 to 0.924] | 0.126 [0.055 to 2.67]
  Day 364 (n=20,23,26,28,27,23) | 0.137 [0.025 to 1.31] | 0.124 [0.025 to 0.53] | 0.105 [0.025 to 0.221] | 0.126 [0.025 to 1.31] | 0.12 [0.025 to 0.287] | 0.124 [0.05 to 0.371]

9. Secondary Outcome: Median Prostate-specific Antigen Levels
Time Frame: Day 0 (Baseline), Days 3, 7, 14, and 364
Population: ITT population
Measure: Median (Full Range); unit: nanogram / milliliter
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
nanogram / milliliter
  Day 0 (Baseline) | 15.2 [2.6 to 332] | 31.5 [3.3 to 1730] | 31.5 [2.6 to 901] | 23.1 [3.6 to 586] | 35.3 [2.4 to 1110] | 32 [2 to 1297]
  Day 3 (n=29,30,28,29,33,28) | 13.7 [2.4 to 207] | 29.9 [3 to 1061] | 27.8 [2 to 443] | 22.2 [2.7 to 503] | 26.3 [1.8 to 928] | 25.2 [1.3 to 945]
  Day 7 (n=30,32,32,30,33,28) | 10.6 [1.9 to 138] | 18.5 [2.4 to 420] | 16.5 [1.8 to 234] | 14.8 [2.4 to 339] | 20.8 [1.5 to 611] | 16.9 [0.9 to 476]
  Day 14 (n=29,31,32,29,33,28) | 7.9 [1 to 69.5] | 10.9 [1.8 to 155] | 9.9 [1.3 to 142] | 7.1 [1.4 to 213] | 13.4 [0.4 to 490] | 8.35 [0.4 to 163]
  Day 364 (n=20,23,26,28,27,22) | 0.45 [0.1 to 5.5] | 0.6 [0.1 to 21.2] | 0.95 [0.1 to 21.6] | 0.9 [0.1 to 135] | 0.8 [0.1 to 48.6] | 0.3 [0.1 to 9.4]

10. Secondary Outcome: Median Values of Di-Hydrotestosterone
Time Frame: Day 0 (Baseline), Days 1, 3, 7, 14, and 364
Population: ITT population
Measure: Median (Full Range); unit: picogram / milliliter
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
picogram / milliliter
  Day 0 (Baseline; n=25,30,26,23,23,25) | 430 [140 to 2600] | 330 [94 to 760] | 310 [170 to 630] | 330 [20 to 760] | 350 [160 to 640] | 290 [160 to 550]
  Day 1 (n=23,27,25,24,26,24) | 130 [41 to 320] | 95 [54 to 290] | 110 [44 to 250] | 130 [30 to 380] | 110 [60 to 480] | 115 [49 to 220]
  Day 3 (n=23,27,25,25,27,25) | 82 [22 to 150] | 67 [32 to 130] | 70 [22 to 130] | 66 [25 to 180] | 73 [10 to 190] | 67 [10 to 180]
  Day 7 (n=26,30,24,26,30,22) | 63 [10 to 260] | 65 [31 to 220] | 61.5 [22 to 150] | 56.5 [21 to 130] | 61 [20 to 240] | 77.5 [20 to 240]
  Day 14 (n=19,27,25,23,25,27) | 68 [10 to 440] | 51 [22 to 120] | 42 [10 to 110] | 57 [10 to 110] | 59 [10 to 130] | 53 [32 to 250]
  Day 364 (n=17,21,20,25,25,21) | 41 [10 to 79] | 39 [10 to 73] | 34 [10 to 72] | 40 [10 to 120] | 39 [10 to 210] | 40 [10 to 130]

11. Secondary Outcome: Median Values for Serum Luteinizing Hormone
Time Frame: Day 0 (Baseline), Days 1, 3, 7, 14, and 364
Population: ITT population
Measure: Median (Full Range); unit: international units / liter
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
international units / liter
  Day 0 (Baseline) | 3.8 [0.5 to 9.6] | 4 [1.6 to 15] | 5.05 [1.2 to 27.6] | 5.6 [1 to 18] | 3.9 [1.6 to 25.9] | 6 [1.6 to 19.5]
  Day 1 (n=28,30,32,28,31,30) | 0.8 [0.05 to 5.7] | 0.65 [0.3 to 3.4] | 0.7 [0.2 to 4.6] | 0.9 [0.2 to 5.8] | 0.7 [0.3 to 7.2] | 0.75 [0.4 to 4.6]
  Day 3 (n=29,30,28,29,33,28) | 0.5 [0.1 to 2.7] | 0.5 [0.2 to 1.9] | 0.5 [0.2 to 2.1] | 0.5 [0.2 to 1.3] | 0.4 [0.2 to 2.4] | 0.55 [0.2 to 1.8]
  Day 7 (n=30,32,32,30,33,28) | 0.7 [0.05 to 5.7] | 0.5 [0.2 to 2.5] | 0.6 [0.2 to 3.4] | 0.5 [0.05 to 3.4] | 0.5 [0.2 to 2.5] | 0.75 [0.2 to 4.3]
  Day 14 (n=29,31,32,29,33,28) | 0.5 [0.05 to 7.4] | 0.3 [0.1 to 2.8] | 0.35 [0.05 to 4.5] | 0.3 [0.05 to 5.1] | 0.3 [0.05 to 1.8] | 0.3 [0.05 to 4.8]
  Day 364 (n=20,23,26,28,27,22) | 0.3 [0.05 to 1.5] | 0.3 [0.05 to 2.3] | 0.2 [0.05 to 0.6] | 0.4 [0.05 to 2.5] | 0.2 [0.05 to 0.8] | 0.3 [0.05 to 1.3]

12. Secondary Outcome: Median Values for Follicle Stimulation Hormone
Time Frame: Day 0 (Baseline), Days 1, 3, 7, 14, and 364
Population: ITT population
Measure: Median (Full Range); unit: international units / liter
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
international units / liter
  Day 0 (Baseline) | 8.35 [2.3 to 45.4] | 9.25 [2.4 to 39.2] | 9 [3.8 to 40.7] | 9.7 [4.1 to 61.7] | 7 [2.3 to 76.1] | 10.2 [1.8 to 67.9]
  Day 1 (n=28,30,32,28,31,30) | 5.15 [1.4 to 28.6] | 5.65 [1.5 to 24.8] | 5.35 [2.3 to 24.8] | 6.2 [2.4 to 46.2] | 4.4 [1.7 to 55.2] | 5.9 [1 to 47.4]
  Day 3 (n=29,30,28,29,33,28) | 2.9 [0.8 to 14.4] | 3.15 [1 to 14.1] | 3.25 [1.2 to 13.5] | 3.3 [1.4 to 9.3] | 2.5 [0.9 to 31.5] | 3.1 [0.7 to 24.1]
  Day 7 (n=30,32,32,30,33,28) | 2.7 [0.3 to 9.3] | 1.95 [0.6 to 12.9] | 1.85 [0.8 to 8.7] | 1.85 [0.7 to 16] | 1.4 [0.5 to 16.1] | 2.55 [0.6 to 13.1]
  Day 14 (n=29,31,32,29,33,28) | 1.6 [0.05 to 11.5] | 1.1 [0.3 to 11.2] | 0.9 [0.2 to 7.9] | 0.8 [0.2 to 8.5] | 0.7 [0.1 to 8] | 0.95 [0.2 to 14.5]
  Day 364 (n=20,23,26,28,27,22) | 1.8 [0.2 to 7] | 1.5 [0.2 to 7.6] | 1.45 [0.2 to 6.4] | 1.75 [0.1 to 13] | 1.1 [0.3 to 5.3] | 2.2 [0.3 to 11.4]

13. Secondary Outcome: The Number of Patients With Abnormal Liver Function Tests
Description: The number of patients who had abnormal (defined as above upper limit of normal range(ULN)) alanine aminotransferase(ALT), aspartate aminotransferase levels, and bilirubin levels. Also includes the number of patients who had ALT increases >3x ULN, and patients with ALT increases >3x ULN with concurrent increases in bilirubin >1.5 ULN.
Time Frame: 364 days
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
participants
  Abnormal alanine aminotransferase (ALT) | 6 | 10 | 15 | 13 | 8 | 9
  Abnormal aspartate aminotransferase | 7 | 10 | 15 | 8 | 13 | 13
  Abnormal bilirubin | 2 | 5 | 1 | 2 | 5 | 1
  ALT >3x ULN | 3 | 8 | 12 | 13 | 7 | 8
  ALT>3x ULN and bilirubin >1.5x ULN | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: The Number of Patients With Markedly Abnormal Changes in Vital Signs or Body Weight
Description: Vital sign and body weight values at the end of the trial are compared to baseline values. The table represents the number of patients in each group with normal baseline values and markedly abnormal end-of-study values.
Time Frame: Day 364
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Number analyzed (Participants) | 30 | 32 | 32 | 30 | 33 | 30
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0 | 0 | 2 | 2 | 2
  Diastolic blood pressure >=105 and increase >=15 | 3 | 3 | 4 | 3 | 0 | 2
  Pulse <=50 and decrease >=15 from baseline | 0 | 2 | 0 | 2 | 1 | 1
  Pulse >=120 and increase of >=15 from baseline | 0 | 0 | 0 | 1 | 0 | 0
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0 | 1 | 0 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 3 | 2 | 4 | 0 | 3 | 2
  Weight decrease of >=7% from baseline | 0 | 1 | 1 | 3 | 1 | 0
  Weight increase of >=7% from baseline | 3 | 4 | 6 | 5 | 4 | 1

ADVERSE EVENTS:
Arm/Group | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Serious Adverse Events (participants affected / at risk) | 3 | 6 | 4 | 4 | 6 | 4
Other Adverse Events (participants affected / at risk) | 17 | 21 | 24 | 19 | 23 | 20
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Anaemia (Blood and lymphatic system disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Acute myocardial infarction (Cardiac disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Angina pectoris (Cardiac disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Angina unstable (Cardiac disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Atrioventricular block complete (Cardiac disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Cardiac failure (Cardiac disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Coronary artery stenosis (Cardiac disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Myocardial infarction (Cardiac disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Supraventricular tachycardia (Cardiac disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Corneal defect (Eye disorders) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Ulcerative keratitis (Eye disorders) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Disease progression (General disorders) | 1/30 (1) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Bronchopneumonia (Infections and infestations) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Gastroenteritis viral (Infections and infestations) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Pneumonia (Infections and infestations) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Alanine aminotransferase increased (Investigations) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Aspartate aminotransferase increased (Investigations) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Blood alkaline phosphatase increased (Investigations) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Gamma-glutamyltransferase increased (Investigations) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Cachexia (Metabolism and nutrition disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/30 (1) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 1/32 (1) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 0/32 (0) | 1/32 (2) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Metastases to penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Cerebrovascular accident (Nervous system disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 2/33 (2) | 0/30 (0)
Ischaemic stroke (Nervous system disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Spinal cord compression (Nervous system disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Depression (Psychiatric disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Suicide attempt (Psychiatric disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Hydronephrosis (Renal and urinary disorders) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Urinary retention (Renal and urinary disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Anuria (Renal and urinary disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Calculus bladder (Renal and urinary disorders) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Haematuria (Renal and urinary disorders) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Ureteric obstruction (Renal and urinary disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Hypertension (Vascular disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 200/80 | Degarelix 200/120 | Degarelix 200/160 | Degarelix 240/80 | Degarelix 240/120 | Degarelix 240/160
Atrial fibrillation (Cardiac disorders) | 0/30 (0) | 1/32 (1) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 2/30 (2)
Atrioventricular block first degree (Cardiac disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 2/30 (2) | 1/33 (1) | 0/30 (0)
Diarrhoea (Gastrointestinal disorders) | 1/30 (2) | 3/32 (4) | 2/30 (2) | 0/30 (0) | 1/33 (1) | 2/30 (2)
Constipation (Gastrointestinal disorders) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 2/30 (2) | 0/33 (0) | 1/30 (1)
Injection site pain (General disorders) | 1/30 (1) | 3/32 (3) | 6/32 (17) | 0/30 (0) | 6/33 (11) | 2/30 (2)
Fatigue (General disorders) | 2/30 (2) | 1/32 (1) | 2/32 (3) | 3/30 (4) | 1/33 (1) | 2/30 (2)
Injection site swelling (General disorders) | 0/30 (0) | 2/32 (4) | 2/32 (7) | 0/30 (0) | 1/33 (3) | 1/30 (1)
Pyrexia (General disorders) | 3/30 (4) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 2/30 (5)
Injection site erythema (General disorders) | 0/30 (0) | 0/32 (0) | 2/32 (2) | 0/30 (0) | 1/33 (1) | 1/30 (1)
Asthenia (General disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 2/33 (2) | 1/30 (1)
Injection site inflammation (General disorders) | 0/30 (0) | 2/32 (2) | 1/32 (1) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Urinary tract infection (Infections and infestations) | 2/30 (2) | 2/32 (2) | 2/32 (4) | 2/30 (2) | 2/33 (2) | 1/30 (1)
Influenza (Infections and infestations) | 1/30 (1) | 0/32 (0) | 2/32 (2) | 0/30 (0) | 1/33 (1) | 2/30 (2)
Nasopharyngitis (Infections and infestations) | 2/30 (3) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 2/33 (2) | 1/30 (1)
Pneumonia (Infections and infestations) | 1/30 (1) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 2/30 (2)
Bronchitis (Infections and infestations) | 0/30 (0) | 0/32 (0) | 2/32 (2) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Weight increase (Investigations) | 1/30 (1) | 3/32 (3) | 4/32 (4) | 4/30 (4) | 3/33 (3) | 2/30 (2)
Alanine aminotransferase increased (Investigations) | 2/30 (2) | 1/32 (1) | 3/32 (4) | 0/30 (0) | 1/33 (3) | 1/30 (1)
Blood alkaline phosphatase increased (Investigations) | 2/30 (2) | 0/32 (0) | 2/32 (3) | 0/30 (0) | 1/33 (1) | 1/30 (1)
Aspartate aminotransferase increased (Investigations) | 1/30 (1) | 0/32 (0) | 2/32 (2) | 0/30 (0) | 1/33 (3) | 1/30 (1)
Blood urea increased (Investigations) | 0/30 (0) | 0/32 (0) | 2/32 (2) | 2/30 (3) | 0/33 (0) | 0/32 (0)
Blood creatinine increased (Investigations) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 2/30 (2) | 0/33 (0) | 0/30 (0)
Weight decreased (Investigations) | 0/30 (0) | 0/32 (0) | 2/32 (2) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/30 (1) | 3/32 (3) | 1/32 (1) | 1/30 (1) | 2/33 (2) | 1/30 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/30 (2) | 0/32 (0) | 2/32 (3) | 0/30 (0) | 0/33 (0) | 2/30 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/30 (0) | 1/32 (1) | 1/32 (2) | 2/30 (3) | 2/33 (2) | 0/30 (0)
Headache (Nervous system disorders) | 0/30 (0) | 0/32 (0) | 2/32 (2) | 2/30 (2) | 0/33 (0) | 2/30 (3)
Syncope vasovagal (Nervous system disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 2/30 (2) | 0/33 (0) | 0/30 (0)
Insomnia (Psychiatric disorders) | 1/30 (1) | 1/32 (1) | 3/32 (3) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Anxiety (Psychiatric disorders) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 1/30 (1) | 2/33 (2) | 1/30 (1)
Haematuria (Renal and urinary disorders) | 0/30 (0) | 0/32 (0) | 2/32 (2) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0/30 (0) | 0/32 (0) | 0/32 (0) | 2/30 (2) | 0/33 (0) | 0/30 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2/30 (2) | 1/32 (1) | 2/32 (2) | 1/30 (1) | 0/33 (0) | 1/30 (1)
Testicular atrophy (Reproductive system and breast disorders) | 2/30 (2) | 0/32 (0) | 1/32 (1) | 0/30 (0) | 1/33 (1) | 0/30 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2/30 (2) | 0/32 (0) | 0/32 (0) | 1/30 (1) | 0/33 (0) | 0/30 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/30 (2) | 1/32 (1) | 2/32 (3) | 1/30 (1) | 0/33 (0) | 3/30 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/30 (0) | 2/32 (3) | 0/32 (0) | 0/30 (0) | 1/33 (1) | 1/30 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/30 (2) | 0/32 (0) | 2/32 (2) | 0/30 (0) | 0/33 (0) | 0/30 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0/30 (0) | 0/32 (0) | 1/32 (1) | 1/30 (1) | 3/33 (3) | 0/30 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/30 (1) | 0/32 (0) | 2/32 (2) | 1/30 (2) | 1/33 (1) | 0/30 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2/30 (2) | 0/32 (0) | 0/32 (0) | 0/30 (0) | 0/33 (0) | 1/30 (1)
Hot flush (Vascular disorders) | 14/30 (16) | 8/32 (8) | 10/32 (13) | 11/30 (14) | 9/33 (9) | 10/30 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.